CLINICAL TRIAL: NCT05410548
Title: Can Comorbidity Screening and Referral by Prosthetists Enhance Post-Amputation Care?
Brief Title: Comorbidity Screening and Referral by Prosthetists
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Delaware (Other)
Collaborators: Independence Prosthetics-Orthotics, Inc. (Unknown); Orthotic and Prosthetic Education and Research Foundation (OPERF) (Other)
Responsible Party: Principal Investigator, Jaclyn Sions, Assistant Professor, University of Delaware
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 1865677
Record Dates: First submitted 2022-06-02; First posted 2022-06-08 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2023-05

CONDITIONS: Limb Ischemia; Low Back Pain; Depression; Neuropathy;Peripheral; Amputation
Keywords: comorbidity; peripheral arterial disease; sensation; back pain; mental health; amputation
MeSH Terms: conditions — Low Back Pain; Depression; Neuritis; Peripheral Arterial Disease; Back Pain; Psychological Well-Being | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Patient participant satisfaction surveys, which are a primary outcome, will be collected in sealed envelopes and data will be entered by a research team member who is not a practitioner conducting the intervention. Satisfaction data will be stored in a separate database that is concealed from practitioners until the last participant completes their 3-month follow-up. Three-month follow-ups will occur remotely and without practitioner input. Patient care minutes will be extracted from the electronic medical record generated during actual patient visits.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard-of-Care (Other): Patient participants will receive routine standardized prosthetic follow-up care by a certified prosthetist, including evaluation of prosthesis use, prosthesis-enabled mobility, socket comfort and sock ply usage, falls, body anthropometrics, and functional mobility.
  Interventions: Other: Standard-of-Care
- Standard-of-Care + Clinical Screening (Experimental): In addition to routine, standardized prosthetic follow-up care, patient participants will receive comorbidity screening for contralateral limb peripheral arterial disease, peripheral neuropathy, major depression, and greater than low risk for persistent low back pain. Participants will be educated on clinical screening findings, provided a copy of their screening results to share with their medical providers, and their results will be securely sent to their primary care provider.
  Interventions: Other: Standard-of-Care; Other: Clinical Screening

INTERVENTIONS:
Other: Standard-of-Care — Participants with a major unilateral transfemoral or transtibial amputation will undergo a standardized medical history and medication review, complete questionnaires evaluating prosthesis use, comfort, and mobility, receive a clinical examination of height, weight and limb circumference, and complete three performance-based mobility outcome measures.
Other: Clinical Screening — Participants will complete the following self-report questionnaires: (a) the Patient Health Questionnaire-9 item, which may suggest major depression and/or suicidal ideation; and (b) the STarT Back Screening Tool, a 6-item tool used to screen for greater than low-risk for persistent, bothersome and disabling low back pain. Prosthetists will perform palpation of the contralateral dorsalis pedis and posterior tibial pulses and note presence or absence, as an indicator of peripheral arterial disease. Prosthetists will evaluate protective sensation of the contralateral foot through Semmes-Weinstein monofilament assessment of the great toe, the 1st and 3rd metatarsal heads. The prosthetist will record the results in a letter that is sent to the patient's primary care provider, and provide a copy of the letter to the patient after discussing the results for each of the screens.
  Arms: Standard-of-Care + Clinical Screening

SUMMARY:
Lower-limb amputation is associated with life-altering and life-limiting comorbidities. Currently, onus is on primary care providers to diagnose, educate, and refer patients for appropriate management. Recently our laboratory has found, however, that of adults post-amputation seen in an outpatient Limb Loss Clinic presenting with comorbidities, >50% are unaware they have signs of peripheral arterial disease and/or neuropathy. Lack of patient awareness and thus, inadequate comorbidity management, may contribute to suboptimal patient outcomes post-amputation. As a first step in this research line, the proposed project will help determine if comorbidity screening by prosthetists during routine care visits for patients post-amputation may enhance comorbidity awareness, increase patient satisfaction in prosthetic services, and reduce gratuitous prosthetic service utilization. During a follow-up visit, seventy patients following a unilateral lower-limb amputation will be randomized into either a standard-of-care group or a standard of-care plus group. The standard-of-care plus group will receive clinical screenings by a certified prosthetist for peripheral arterial disease, peripheral neuropathy, depression, and high-risk for persistent back pain; patient education on findings; and each participant's primary care provider will receive screening results. The long-term goal of this research is to determine if prosthetists can maximize their utility in an interdisciplinary care team, while enhancing patient outcomes post-amputation.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking and -reading
* Unilateral transtibial (i.e., below-knee) or transfemoral (i.e., above-knee) amputation
* Utilization of a prosthesis for at least 1 year
* Willingness to have screening results communicated to their primary care provider
* Receiving prosthetic care at Independence Prosthetics-Orthotics, Inc.

Exclusion Criteria:

* Cognitive impairment precluding ability to consent to study participation
* Contralateral limb amputation greater than toe-level
* Severe vision or hearing loss
* Receipt of a replacement prosthetic component within the 3 months prior to study enrollment
* Hospitalization within the 3 months prior to study enrollment

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2022-06-09 (Actual); Primary Completion 2023-01-30 (Actual); Study Completion 2023-01-30 (Actual)

PRIMARY OUTCOMES:
Orthotic and Prosthetic Limb User Survey of Mobility (OPUS): Satisfaction with Device and Services | 3-month follow-up
  This questionnaire evaluates device function, fit, and cosmesis, as well as education, timeliness, and courtesy of the practitioner through 21 items. Items are scored on a 5-point Likert scale and higher scores indicate greater satisfaction. Items 1-11 are summed for the Satisfaction with Device subscale score (range: 11-55) and items 12-21 are summed for the Satisfaction with Services subscale score (range: 10-50).
Client Satisfaction Inventory-short form | 3-month follow-up
  This 9-item survey assesses how the individual feels about the services they have received. Items are rated from 1 (none of the time) to 7 (all of the time) and summed for a total possible score of 7-63. Higher scores indicate greater satisfaction.
Prosthetic service utilization | through study completion, an average of 3 months
  Number of patient care minutes extracted from each participant's electronic medical record

CONTACTS AND LOCATIONS:
Overall Officials: Jaclyn M Sions, PhD, DPT, Principal Investigator — University of Delaware
Locations (1):
- University of Delaware STAR Campus, Newark, Delaware, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified patient participant data are available from the corresponding author upon reasonable request and with completion of a data use agreement to protect participant confidentiality.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Individual patient participant data that underlie results will be available beginning 3 months following publication of the primary results and ending 5 years following publication of the primary results to researchers who provide a methodologically sound proposal and complete a data sharing agreement.
Access Criteria: Proposals should be directed to J. Megan Sions, PT, DPT, PhD, the study's principal investigator, in writing at megsions@udel.edu. To gain access to individual patient participant data, requestors will need to sign a data access agreement with the principal investigator's home institution, i.e., the University of Delaware.

DOCUMENTS (1):
  • Informed Consent Form (2022-03-28): https://cdn.clinicaltrials.gov/large-docs/48/NCT05410548/ICF_000.pdf